CLINICAL TRIAL: NCT02408471
Title: Post-Approval Study Protocol; Ascension® MCP Finger Implant; PyroCarbon Metacarpophalangeal Total Joint Prosthesis
Brief Title: Ascension® Post- Approval Study; PyroCarbon Metacarpophalangeal Total Joint Prosthesis
Acronym: MCP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Priorities
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MCP-002; NCT01398735 (obsolete NCT alias)
Record Dates: First submitted 2014-11-04; First posted 2015-04-03 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus; Osteoarthritis; Post-traumatic Arthritis
Keywords: Arthritis; Rheumatoid Arthritis; Systemic Lupus Erythematosus; Osteoarthritis; Autoimmune Diseases; Connective Tissue Diseases; Immune System Diseases; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Osteoarthritis; Arthritis; Autoimmune Diseases; Connective Tissue Diseases; Immune System Diseases; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ascension® MCP Finger Implant (Other): Single arm study, patient treated with Ascension® PyroCarbon MCP implant.
  Interventions: Device: Ascension® MCP Finger Implant

INTERVENTIONS:
Device: Ascension® MCP Finger Implant — Patients who meet inclusion/ exclusion criteria are treated with the Ascension® MCP.

SUMMARY:
This study is a non-randomized, consecutive enrollment, one-year post-approval study of patients who are treated with the Ascension® MCP.

ELIGIBILITY:
Inclusion Criteria:

* Indications consistent with the FDA approved Indications For Use: Index, long, ring, or small finger metacarpophalangeal (MCP) joints that exhibit symptoms of pain, limited motion, or inadequate bony alignment (i.e., subluxation/dislocation) secondary to articular destruction or degenerative disease related to rheumatoid arthritis, systemic lupus erythematosus, osteoarthritis, or post-traumatic arthritis where soft tissue reconstruction can provide adequate stabilization
* Willing to participate in the study
* Signed an Informed Consent Form
* The means and ability to return for all required study visits
* Are not transient

Exclusion Criteria:

Patients who have any of the following contraindications will be excluded from the study:

* Inadequate bone stock at the implantation site
* Active infection in the MCP joint
* Nonfunctioning and irreparable MCP musculotendinous system
* Physical interference with or by other prostheses during implantation or use
* Procedures requiring modification of the prosthesis
* Skin, bone, circulatory and/or neurological deficiency at the implantation site

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2002-06 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tummon, Study Director — Sponsor- Integra LifeSciences
Locations (9):
- United States (9):
  - Southwest Shoulder Elbow and Hand Center, P.C., Tucson, Arizona
  - Bloomington Bone and Joint Clinic, Bloomington, Indiana
  - Reconstructive Hand Surgeons of Indiana, Carmel, Indiana
  - The Indiana Hand Center, Indianapolis, Indiana
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The Center for Ortho/ Neuro Care & Research, Bend, Oregon
  - ROC Houston, PA, Houston, Texas
  - Fondren Orthopedic Group, L.L.P., Houston, Texas
  - The Hand Center of San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from 25 June 2002 to early termination on 03 January 2015.
Pre-assignment Details: One bilateral participant completed the study in 2010 for the left hand and the same participant enrolled in the study again in 2011 for the right hand. Each enrollment is accounted for separately as appropriate for the total number of participants enrolled.
Period: Overall Study
Arm/Group | Ascension® MCP Finger Implant
Started | 97
Completed | 69
Not Completed | 28

BASELINE CHARACTERISTICS:
Population: One bilateral participant enrolled in the study twice. The second enrollment was the contralateral hand after this participant completed the study.
Units Other Than Participants: hands
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
Number analyzed (hands) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only data available for age used for analysis.
  years
    number analyzed (Participants) | 92
    (all) | 59.9 (12.0)
Sex: Female, Male [Count of Units; unit: hands]
  Female | 48
  Male | 49
Race/Ethnicity, Customized [Count of Units; unit: hands] — Unknown indicates queried data that returned nothing recorded on medical charts. 46 participants' information (47 hands) could not be retrieved due to site closure.
  hands
    Race/Ethnicity: Black | 1
    Race/Ethnicity: Caucasian/White | 42
    Race/Ethnicity: Hispanic/Latino | 1
    Race/Ethnicity: Unknown | 6
    Race/Ethnicity: Not Retrieved | 47
Region of Enrollment [Number; unit: participants]
  United States | 97
Number of Affected Joints [Number; unit: joints] | 162

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Revisions
Description: Count of participants with a revision surgery.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
Participants | 6

2. Secondary Outcome: Change in Joint Range of Motion
Description: Range of motion measured by clinical assessment for joint extension and joint flexion. Measurements of extension and flexion made and recorded to the nearest degree using a goniometer with the wrist in the neutral position. Extension measured with fingers actively extended and flexion measured after the participant made a fist.
Time Frame: Preoperatively to 12 months
Population: Number of Participants Analyzed indicates overall population throughout the given time frame with any available joint data necessary for the assessment specified.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: joints
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
Number analyzed (joints) | 122
degrees
  Joint Extension: number analyzed (joints) | 115
  Joint Extension | 18.2 (30.2)
  Joint Flexion | -6.2 (25.8)

3. Secondary Outcome: Change in Radial-Ulnar Deviation
Description: Measurements of ulnar deviation made for each implanted metacarpophalangeal (MCP) joint. Measurements made to the nearest degree using a goniometer with the participant's wrist in a neutral position and the finger(s) fully extended (e.g., no extension deficit). Radial deviation or ulnar deviation direction checked.
Time Frame: Preoperatively to 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: joints
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
Number analyzed (joints) | 102
degrees
  Radial Deviation: number analyzed (Participants) | 1
  Radial Deviation: number analyzed (joints) | 1
  Radial Deviation | 0 (NA) — Standard Deviation could not be calculated due to insufficient participant data available for Radial Deviation.
  Ulnar Deviation | -9.4 (21.1)

4. Secondary Outcome: Change in Tip Pinch
Description: Quantitative measurements of opposition tip pinch strength was made for each implanted digit. Measurements made using a pinch meter.
  For each strength measurement, the participant made 3 attempts with the maximum value recorded.
  If the participant could not perform the pinch test due to inflammation, excessive pain, or some other reason, DNA (which stands for "Did Not Attempt") was recorded. If the participant performs the pinch test but cannot register significant load, the value zero (0) was recorded.
Time Frame: Preoperatively to 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms
Units Other Than Participants: joints
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
Number analyzed (joints) | 113
kilograms | 1.3 (1.9)

5. Secondary Outcome: Change in Grip Strength
Description: Implanted hand grip strength measured using a grip dynamometer instrument.
Time Frame: Preoperatively to 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms
Units Other Than Participants: joints
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
Number analyzed (joints) | 108
kilograms | -0.8 (14.8)

6. Secondary Outcome: Function Visual Analog Scale (VAS)
Description: VAS Function based on a scale of 0 to 100 as completed by the participant with 0 indicating worse function and 100 indicating normal function
Time Frame: Preoperatively, 6 weeks, 12 weeks, 6 months, and 12 months
Population: Participants with available data necessary for the assessment specified for the given time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
score on a scale
  Preoperatively | 29.7 (20.6)
  6 Weeks: number analyzed (Participants) | 89
  6 Weeks | 52.7 (25.9)
  12 Weeks: number analyzed (Participants) | 88
  12 Weeks | 70.9 (25.2)
  6 Months: number analyzed (Participants) | 71
  6 Months | 75.2 (25.7)
  12 Months: number analyzed (Participants) | 68
  12 Months | 83.2 (17.7)

7. Secondary Outcome: Joint Pain Visual Analog Score (VAS)
Description: VAS Joint Pain based on a scale of 0 to 100 as completed by the participant with 0 indicating no pain and 100 indicating severe pain.
Time Frame: Preoperatively, 6 Weeks, 12 Weeks, 6 Months, 12 Months
Population: Participants with available data necessary for the assessment specified for the given time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
score on a scale
  Preoperatively | 65.3 (28.4)
  6 Weeks: number analyzed (Participants) | 89
  6 Weeks | 16.0 (20.0)
  12 Weeks: number analyzed (Participants) | 88
  12 Weeks | 11.3 (18.8)
  6 Months: number analyzed (Participants) | 69
  6 Months | 10.5 (20.5)
  12 Months: number analyzed (Participants) | 69
  12 Months | 11.8 (19.4)

8. Secondary Outcome: Cosmetic Appearance Visual Analog Scale (VAS)
Description: VAS Cosmetic Appearance based on a scale of 0 to 100 as completed by the participant with 0 indicating worst appearance and 100 indicating normal appearance.
Time Frame: Preoperatively, 6 Weeks, 12 Weeks, 6 Months, and 12 months
Population: Participants with available data necessary for the assessment specified for the given time frame.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
score on a scale
  Preoperatively | 39.8 (33.8)
  6 Weeks: number analyzed (Participants) | 89
  6 Weeks | 71.1 (23.8)
  12 Weeks: number analyzed (Participants) | 88
  12 Weeks | 75.4 (25.4)
  6 Months: number analyzed (Participants) | 71
  6 Months | 78.1 (25.5)
  12 Months: number analyzed (Participants) | 68
  12 Months | 83.0 (25.6)

9. Secondary Outcome: Joint Position
Description: Joint position for the affected finger determined by radiographic evaluation. Standard anteroposterior (AP), oblique, and lateral radiographs were made at the pre-operative and all post-operative evaluation visits of the hand(s) in which the Ascension MCP device was implanted. Joint position was classified as reduced, subluxed, dislocated, or (data) missing.
Time Frame: Preoperatively, 6 weeks, 12 weeks, 6 months, and 12 months
Population: Number analyzed for each specified time frame and category includes participants with available finger data.
Measure: Count of Units; unit: fingers
Units Other Than Participants: fingers
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 97
Number analyzed (fingers) | 161
fingers
  Preoperatively: Reduced | 78
  Preoperatively: Subluxed | 62
  Preoperatively: Dislocated | 20
  Preoperatively: Missing | 1
  6 Weeks: number analyzed (Participants) | 93
  6 Weeks: number analyzed (fingers) | 155
  6 Weeks: Reduced | 152
  6 Weeks: Subluxed | 0
  6 Weeks: Dislocated | 2
  6 Weeks: Missing | 1
  12 Weeks: number analyzed (Participants) | 89
  12 Weeks: number analyzed (fingers) | 152
  12 Weeks: Reduced | 148
  12 Weeks: Subluxed | 2
  12 Weeks: Dislocated | 0
  12 Weeks: Missing | 2
  6 Months: number analyzed (Participants) | 74
  6 Months: number analyzed (fingers) | 131
  6 Months: Reduced | 122
  6 Months: Subluxed | 2
  6 Months: Dislocated | 1
  6 Months: Missing | 6
  12 Months: number analyzed (Participants) | 69
  12 Months: number analyzed (fingers) | 123
  12 Months: Reduced | 118
  12 Months: Subluxed | 3
  12 Months: Dislocated | 0
  12 Months: Missing | 2

10. Secondary Outcome: Component Migration
Description: Component migration determined by radiographic assessment. Migration of the device was classified as none, yes, or (data) missing.
Time Frame: 6 Weeks, 12 Weeks, 6 Months, 12 Months
Population: Number analyzed for each specified time frame and category includes participants with available implanted device data.
Measure: Count of Units; unit: devices
Units Other Than Participants: devices
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 93
Number analyzed (devices) | 155
devices
  6 Weeks: None | 155
  6 Weeks: Yes | 0
  6 Weeks: Missing | 0
  12 Weeks: number analyzed (Participants) | 89
  12 Weeks: number analyzed (devices) | 152
  12 Weeks: None | 151
  12 Weeks: Yes | 0
  12 Weeks: Missing | 1
  6 Months: number analyzed (Participants) | 74
  6 Months: number analyzed (devices) | 131
  6 Months: None | 130
  6 Months: Yes | 1
  6 Months: Missing | 0
  12 Months: number analyzed (Participants) | 69
  12 Months: number analyzed (devices) | 123
  12 Months: None | 123
  12 Months: Yes | 0
  12 Months: Missing | 0

11. Secondary Outcome: Bone Changes by Device
Description: X-rays were examined to determine if the implant components demonstrate stable fixation in the bone. Bone changes were classified as no changes (i.e., none), any bone changes, or (data) missing.
Time Frame: 6 Weeks, 12 Weeks, 6 Months, 12 Months
Population: Number analyzed for each specified time frame and category includes participants with available finger data.
Measure: Count of Units; unit: devices
Units Other Than Participants: devices
Arm/Group | Ascension® MCP Finger Implant
Number analyzed (Participants) | 93
Number analyzed (devices) | 155
devices
  6 Weeks: None | 154
  6 Weeks: Any Bone Changes | 1
  6 Weeks: Missing | 0
  12 Weeks: number analyzed (Participants) | 89
  12 Weeks: number analyzed (devices) | 152
  12 Weeks: None | 148
  12 Weeks: Any Bone Changes | 3
  12 Weeks: Missing | 1
  6 Months: number analyzed (Participants) | 74
  6 Months: number analyzed (devices) | 131
  6 Months: None | 103
  6 Months: Any Bone Changes | 28
  6 Months: Missing | 0
  12 Months: number analyzed (Participants) | 69
  12 Months: number analyzed (devices) | 123
  12 Months: None | 68
  12 Months: Any Bone Changes | 52
  12 Months: Missing | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to study completion or termination, up to 1 year.
Description: Adverse events were recorded on the appropriate Case Report Form. The investigator would inform the sponsor within 24 hours in the event of:
  * A severe, unexpected, device related complication or adverse event; or
  * A re-operation procedure for device removal or additional soft-tissue reconstruction.
Arm/Group | Ascension® MCP Finger Implant
All-Cause Mortality (participants affected / at risk) | 0/97
Serious Adverse Events (participants affected / at risk) | 25/97
Other Adverse Events (participants affected / at risk) | 30/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ascension® MCP Finger Implant (N=97)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Deformity (Musculoskeletal and connective tissue disorders) | 1 — Possibly related to device
Deformity (Musculoskeletal and connective tissue disorders) | 1
Deformity - Boutonniere (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Deformity - Swan Neck (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
DIP Mallet (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
DIP pin removal (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Dislocation (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
Dislocation (Musculoskeletal and connective tissue disorders) | 1 — Possibly related to device
Emergent Prostate Surgery (Renal and urinary disorders) | 1 — Unrelated to device
Excessive Pain (General disorders) | 1 — Unrelated to device
Flexion Contracture (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
Flexion Contracture (Musculoskeletal and connective tissue disorders) | 1
Flexion Contracture, tendon adhesion (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Gastrointestinal (Gastrointestinal disorders) | 1 — Unrelated to device
Increased Stiffness (Musculoskeletal and connective tissue disorders) | 1 — Possibly related to device
Increased Stiffness (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Increased Stiffness (Musculoskeletal and connective tissue disorders) | 1
Loss of Motion (Musculoskeletal and connective tissue disorders) | 1 — Device related
Numbness/Nerve Symptoms (Nervous system disorders) | 1 — Unrelated to device
OA Contralateral Hand (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
OA w/ midcarpal instability (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Osteoarthritis w/ midcarpal instability (Musculoskeletal and connective tissue disorders) | 1 — Possibly related to device
Pain (General disorders) | 1 — Unrelated to device
Pin Protrusion (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Pin Removal (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
PIP Deformities (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Recurrent Radial Deviation (Musculoskeletal and connective tissue disorders) | 1 — Possibly related to device
Recurrent Ulnar Deviation (Musculoskeletal and connective tissue disorders) | 3 — Unrelated to device
Recurrent Ulnar Deviation (Musculoskeletal and connective tissue disorders) | 1 — Possibly related to device
Recurrent Ulnar Deviation (Musculoskeletal and connective tissue disorders) | 1 — Device related
Reduction/Loss of Motion (Musculoskeletal and connective tissue disorders) | 1 — Possibly related to device
Removal of Kirschner wires (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Rupture (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Stiffness (Musculoskeletal and connective tissue disorders) | 3 — Unrelated to device
Stiffness (Musculoskeletal and connective tissue disorders) | 1 — Possibly related to device
Stiffness (Musculoskeletal and connective tissue disorders) | 1 — Device related
Subluxation (Musculoskeletal and connective tissue disorders) | 2 — Possibly related to device
Subluxation (Musculoskeletal and connective tissue disorders) | 1 — Device related
Subluxation (Musculoskeletal and connective tissue disorders) | 1
Subluxation (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Surgery on other hand (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Synovitis/Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 — Possibly related to device
Tendon Adhesion (Musculoskeletal and connective tissue disorders) | 3 — Unrelated to device
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 1 — Unrelated to device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ascension® MCP Finger Implant (N=97)
Back Surgery (Musculoskeletal and connective tissue disorders) | 1
Blistering at tourniquet site (General disorders) | 1
Bone Fracture (Musculoskeletal and connective tissue disorders) | 1 — Possibly device related
Bone Fracture (Musculoskeletal and connective tissue disorders) | 1 — Device Related
Bone Fracture (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
Calcification PIP joint (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Cardiovascular (Cardiac disorders) | 1
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
Clicking, popping, pain in right middle finger (Musculoskeletal and connective tissue disorders) | 1 — Possibly device related
Deformity (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Dislocation (Musculoskeletal and connective tissue disorders) | 1
Excessive Pain (Musculoskeletal and connective tissue disorders) | 1 — Device Related
Excessive Pain (Musculoskeletal and connective tissue disorders) | 1 — Possibly device related
Excessive Swelling (General disorders) | 3 — Unrelated to device
Excessive Swelling (Musculoskeletal and connective tissue disorders) | 1 — Possibly device related
Extension lag (Musculoskeletal and connective tissue disorders) | 1 — Possibly device related
Flexion Contracture (Musculoskeletal and connective tissue disorders) | 1 — Possibly device related
Gastrointestinal-Hospitalized for GI Bleed (Gastrointestinal disorders) | 1
Increased Stiffness (Musculoskeletal and connective tissue disorders) | 2 — Possibly device related
Increased Stiffness (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Infection - superficial (Infections and infestations) | 2 — Unrelated to device
Lacerated EPB tendon (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Legionella infection (Infections and infestations) | 1 — Unrelated to device
Mild, clicking, popping, left index finger (Musculoskeletal and connective tissue disorders) | 1 — Possibly device related
Numbness/Nerve Symptoms (Nervous system disorders) | 1 — Unrelated to device
Pain (General disorders) | 1 — Unrelated to device
Pain Onset (General disorders) | 1 — Unrelated to device
Pin Protrusion (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Pin removal (L) Hand (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
PIP Revision surgery (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Recureent Radial/Ulnar Deviation (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Recurrent Ulnar Deviation (Musculoskeletal and connective tissue disorders) | 1 — Possibly device related
Recurrent Ulnar Deviation (Musculoskeletal and connective tissue disorders) | 2 — Unrelated to device
Recurrent Ulnar Deviation (Musculoskeletal and connective tissue disorders) | 1
Reduction/loss of motion (Musculoskeletal and connective tissue disorders) | 1 — Possibly device related
Revision to another PyroCarbon MCP (Musculoskeletal and connective tissue disorders) | 1
Ring & Small claw deformity (Musculoskeletal and connective tissue disorders) | 1 — Device Related
Scar Adhesion (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
squeaking implant (Injury, poisoning and procedural complications) | 1 — Device Related
Stiffness in Left small finger (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Synovitis (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Tendon Rupture (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device
Total Knee Replacement (Musculoskeletal and connective tissue disorders) | 1
Triggerfinger RR (Musculoskeletal and connective tissue disorders) | 1 — Unrelated to device

LIMITATIONS AND CAVEATS:
Study early terminated by Integra LifeSciences due to poor follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes